CLINICAL TRIAL: NCT06400771
Title: Exploratory, Single-dose, Phase I Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of DNP007 in Healthy Subjects
Brief Title: Safety of DNP007 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Nam-Joon Yi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2402-083-1512
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Liver Transplant Rejection; Liver Transplant; Complications; Steatohepatitis, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 mg/kg (Experimental): 1 mg/kg (IV administered over 30 minutes)
  Interventions: Drug: DNP007
- 2 mg/kg (Experimental): 2 mg/kg (IV administered over 30 minutes)
  Interventions: Drug: DNP007
- 4 mg/kg (Experimental): 4 mg/kg (IV administered over 30 minutes)
  Interventions: Drug: DNP007
- 8 mg/kg (Experimental): 8 mg/kg (IV administered over 30 minutes)
  Interventions: Drug: DNP007

INTERVENTIONS:
Drug: DNP007 — DNP007 is a therapeutic agent that can replace calcineurin inhibitor (CNI), which is a representative factor that can be used as an adhesive for extrahepatic long-term survival patches such as after liver transplantation in patients with liver disease and hepatocellular carcinoma, adult metabolic status, neoplasms, etc. , an anti-ICAM-1 mouse monoclonal minority, is a humanized Fab region that humanizes MD-3 and the Fc region of human IgG1, separated by translational engineering.
  Other Names: MD3, Anti-ICAM1

SUMMARY:
This clinical trial evaluated the safety, tolerability, pharmacokinetic properties, and immunogenicity of DNP007 when administered as a single dose. Since this is a phase 1 study for exploratory evaluation, to the extent that it meets the study objectives, In order to proceed with the minimum number of subjects, a total of 12 people, 3 for each dose group, was planned as the target number.

DETAILED DESCRIPTION:
For volunteers only, screening tests such as questionnaires, physical examinations, and clinical laboratory tests will be conducted within 4 weeks (-28d to -1d) from the date of clinical trial conduct to select test subjects deemed suitable for this clinical trial. Subjects determined to be suitable for this clinical trial are admitted to the Seoul National University Hospital Clinical Trial Center in the afternoon one day (-1d) before the first administration of the investigational drug and must fast for at least 10 hours. In the morning of Day 1, test subjects receive intravenous administration of the clinical trial drug for 30 minutes. Pharmacokinetics, immunogenicity and safety evaluations are conducted according to the planned schedule. Test subjects are hospitalized at the clinical trial center for 4 days (discharged on the 4th day), and after administration of the investigational drug, on 8d, 11d, 15d, 22d (±1d), and 29d (±2d), for pharmacokinetics, immunogenicity, and safety evaluation. Visit the clinical trial center. It proceeds sequentially starting from the lowest dose group, and whether to proceed to the next dose is decided based on the tolerability and safety results up to 15 days of the previous dose.

ELIGIBILITY:
Inclusion Criteria:

* A person whose weight at the time of the screening test is between 50.0 kg and 95 kg and whose body mass index (BMI) is between 18.0 kg/m2 and 30.0 kg/m2
* After receiving sufficient explanation and fully understanding this clinical trial, I voluntarily decided to participate. A person who has made a decision and agreed in writing to follow the precautions
* This test is determined by the examiner through physical examination, clinical laboratory tests, and questionnaires. Persons suitable as test subjects

Exclusion Criteria:

* Clinically significant hepatobiliary system (severe liver failure, viral hepatitis, etc.), kidney (severe renal impairment, etc.), nervous system, immune system, respiratory system, endocrine system, blood/tumor, cardiovascular system (heart failure, etc.), urinary system, Those who have or have a history of mental illness (mood disorder, obsessive-compulsive disorder, etc.), sexual dysfunction, etc
* Persons with a history of gastrointestinal disease (Crohn's disease, ulcer, gastritis, stomach cramps, gastroesophageal reflux disease, etc.) or surgery (excluding simple appendectomy or hernia surgery) that may affect the safety evaluation of clinical investigational drugs
* Persons with a history of related allergy or hypersensitivity (including allergy to aspirin, antibiotics, vaccines, test drugs or their excipients)
* C-reactive protein (CRP) and erythrocyte sedimentation rate in screening tests (ESR) exceeds 1.5 times the upper limit of normal range
* Those with positive serological test results (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test
* A person who has developed an infection or disease within 7 days prior to the first administration of the investigational drug ("disease" refers to an acute [severe or non-severe] condition [e.g., influenza or common cold, etc.])
* Those who have a history of drug abuse or who have tested positive for drugs of abuse in a urine drug screening test
* A person who has taken any prescription drug or herbal medicine within 2 weeks before the scheduled date of first administration of the investigational drug, or who has taken any over-the-counter drug (OTC drug) or health functional food or vitamin preparation including liver function supplements within 1 week (however, the investigator's Depending on the judgment, if other conditions are reasonable, you can be selected as a test subject) or a person who is expected to take the drug
* Clinical trial drugs, barbiturates, etc. within 1 month before the first scheduled administration date. People who have taken drugs that induce drug-metabolizing enzymes or inhibit drug-metabolizing enzymes such as clarithromycin
* Those who consumed grapefruit-containing foods such as grapefruit (grapefruit) or grapefruit juice from 3 days before the first scheduled administration of the investigational drug until the last discharge, and those who cannot refrain from consuming foods containing grapefruit (grapefruit) during the above period
* Those who have unusual eating habits (e.g. drinking more than 1L of grapefruit juice per day) or who are unable to consume the standardized diet provided by the clinical trial center during hospitalization
* Smokers (However, if you quit smoking 3 months or more before the scheduled date of first administration of the investigational drug, you can be selected as a test subject)
* Those who continuously drink alcohol (exceeding 21 units/week, 1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking from 3 days before the first scheduled administration of the investigational drug until the last discharge
* Continuously consumed excessive caffeine (more than 5 units/day) or consumed caffeine-containing foods (coffee, tea (black tea, green tea, etc.), carbonated beverages, coffee milk, nutritional supplements) during the period from 3 days before the first scheduled administration of the investigational drug until the last discharge. Those who cannot refrain from consuming tonic drinks, sports drinks, etc
* A person who received an investigational drug by participating in another clinical trial (including a bioequivalence test) within 6 months before the scheduled date of first administration of the investigational drug
* A person who has donated whole blood or component blood within 1 month within 2 months before the scheduled date of first administration of an investigational drug, or has received a blood transfusion
* Those who are unable or unwilling to use a medically acceptable contraceptive method for themselves or their spouse (or partner) during the period before the clinical trial and at least 4 weeks after the last administration of the investigational drug, and those who do not agree not to donate sperm during that period
* Other persons judged by the investigator to be unsuitable for participation in clinical trials

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0minute (before single intravenous administration), 10, 20, 30 minutes after administration (at completion of infusion), 1, 2, 4, 8, 12, 24, 48, 72, 168hours (Day8), 240hours (Day11), 336hours (Day15), 504hours (Day22±Day1), 672hours (Day29±Day2)
  Pharmacokinetic evaluation variables
The area under the curve up to the last quantifiable time-point (AUClast) | 0minute (before single intravenous administration), 10, 20, 30 minutes after administration (at completion of infusion), 1, 2, 4, 8, 12, 24, 48, 72, 168hours (Day8), 240hours (Day11), 336hours (Day15), 504hours (Day22±Day1), 672hours (Day29±Day2)
  Pharmacokinetic evaluation variables
The area from time of dosing extrapolated to infinity (AUCinf) | 0minute (before single intravenous administration), 10, 20, 30 minutes after administration (at completion of infusion), 1, 2, 4, 8, 12, 24, 48, 72, 168hours (Day8), 240hours (Day11), 336hours (Day15), 504hours (Day22±Day1), 672hours (Day29±Day2)
  Pharmacokinetic evaluation variables
Time to maximum observed plasma concentration (Tmax) | 0minute (before single intravenous administration), 10, 20, 30 minutes after administration (at completion of infusion), 1, 2, 4, 8, 12, 24, 48, 72, 168hours (Day8), 240hours (Day11), 336hours (Day15), 504hours (Day22±Day1), 672hours (Day29±Day2)
  Pharmacokinetic evaluation variables
Half-life (t1/2) | 0minute (before single intravenous administration), 10, 20, 30 minutes after administration (at completion of infusion), 1, 2, 4, 8, 12, 24, 48, 72, 168hours (Day8), 240hours (Day11), 336hours (Day15), 504hours (Day22±Day1), 672hours (Day29±Day2)
  Pharmacokinetic evaluation variables
Oral clearance (CL/F) | 0minute (before single intravenous administration), 10, 20, 30 minutes after administration (at completion of infusion), 1, 2, 4, 8, 12, 24, 48, 72, 168hours (Day8), 240hours (Day11), 336hours (Day15), 504hours (Day22±Day1), 672hours (Day29±Day2)
  Pharmacokinetic evaluation variables
Terminal elimination phase following extravascular (Vz/F) | 0minute (before single intravenous administration), 10, 20, 30 minutes after administration (at completion of infusion), 1, 2, 4, 8, 12, 24, 48, 72, 168hours (Day8), 240hours (Day11), 336hours (Day15), 504hours (Day22±Day1), 672hours (Day29±Day2)
  Pharmacokinetic evaluation variables
Anti-drug antibody measurement (ADA) | 0hour (before administration), 336hours (Day15), and 672hours (Day29±Day2)
  To check the presence or absence of anti-drug antibody expression

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Joon Yi, M.D., Ph.D., Principal Investigator — Department of Surgery, Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hong SK, Han D, Lee SK, Kim J, Hwang ES, Kim H, Lee JI, Hong K, Han ES, Cho JH, Lee JM, Choi Y, Lee KW, Yi NJ, Yang J, Suh KS. Short-term therapy with anti-ICAM-1 monoclonal antibody induced long-term liver allograft survival in nonhuman primates. Am J Transplant. 2021 Sep;21(9):2978-2991. doi: 10.1111/ajt.16486. Epub 2021 Feb 8. PMID 33423374
- [Background] Han DK, Hong SK, Yun IH, Yan JJ, Park J, Kim SW, Seok SH, Kim H, Ji G, Choi Y, Lee KW, Suh KS, Yang J, Yi NJ. Anti-intercellular adhesion molecule 1 monomaintenance therapy induced long-term liver allograft survival without chronic rejection. Am J Transplant. 2024 Oct;24(10):1772-1783. doi: 10.1016/j.ajt.2024.03.037. Epub 2024 Mar 30. PMID 38561059